CLINICAL TRIAL: NCT04656951
Title: Daratumumab for First Line Treatment of Transplant-ineligible Myeloma Patients Followed by Daratumumab Re-treatment at First Relapse
Acronym: GMMG-DADA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Principal Investigator, Christoph Scheid, Principal Investigator, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-3946
Record Dates: First submitted 2020-11-26; First posted 2020-12-07 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab added to VCd in induction, Vd in maintenance and Rd at relapse (Experimental): Daratumumab at standard dose of 1800 mg will be administered subcutaneously at weekly intervals in cycles 1-2 and every 2 weeks in cycles 3-6 and every 4 weeks in cycles 7-8 together with VCD using bortezomib weekly s.c. for 8 cycles of 28 days each, cyclophosphamide i.v. at 500 mg/m2 on d1 of every cycle and dexamethasone p.o. at 20 mg per week.
  Maintenance will be daratumumab subcutaneously every 4 weeks with bortezomib s.c. and dexamethasone 20 mg every 2 weeks until progression or intolerance.
  At relapse/progression treatment will be daratumumab 1800 mg subcutaneously weekly during cycle 1-2, every 2 weeks in cycle 3-6 and every 4 weeks thereafter together with lenalidomide 25 mg p.o. day 1-21 and dexamethasone 20-40 mg weekly.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab added to induction regimen of bortezomib, cyclophosphamide and dexamethasone (VCD), to bortezomib and dexamethasone during maintenance and to lenalidomide and dexamethasone at progression/relapse.
  Other Names: Darzalex

SUMMARY:
Daratumumab for first line treatment of transplant-ineligible myeloma patients followed by daratumumab re-treatment at first relapse (GMMG-DADA)

DETAILED DESCRIPTION:
The aim of the study is to investigate the safety and efficacy of daratumumab added to a standard induction regimen of bortezomib, cyclophosphamide and dexamethasone (VCD). A secondary aim is to assess the efficacy of maintenance therapy until progression using daratumumab in combination with bortezomib and dexamethasone. Thirdly the efficacy of a daratumumab-containing regimen at first relapse shall be tested following a daratumumab-containing first line regimen.

Rationale:

VCD has been established as a standard of care for first line therapy of transplant-eligible patients in Germany. The favorable toxicity profile makes this regimen also suitable for transplant-ineligible patients. Daratumumab has shown to be safe and efficacious in a variety of combinations such as with VMP, Vd or Rd. Using a reduced dose of cyclophosphamide the study shall investigate safety and efficacy of Dara-VCD in the transplant-ineligible patient population.

Maintenance therapy has become standard of care in transplant-eligible and non-eligible patients. However, there is uncertainty whether a single agent maintenance is sufficient or whether a combination therapy is necessary. In this study the safety and efficacy of maintenance with daratumumab in combination with bortezomib and dexamethasone will be assessd with a focus on MRD negativity as a novel endpoint.

The multitude of treatment options at first relapse has generated the need to find an optimal sequence of therapy regimens in first and second line. In particular it is unclear whether the efficacy of daratumumab at relapse is affected by its prior use as part of the first line treatment. Patients in this study will relapse on or after a daratumumab-containing maintenance and shall receive DRd at first relapse. In the POLLUX study patients received DRd but had no prior exposure to daratumumab. Therefore, patients included into the POLLUX study can serve as an indirect control cohort for the present study. If in the present study the PFS after DRd is similar to the PFS of the comparable cohort from the POLLUX study, the assumption is supported that prior exposure to daratumumab does not impair the activity of a subsequent daratumumab-containing regimen at relapse. In addition, the overall efficacy of the whole protocol treatment will be assessed by analyzing PFS2 after relapse from study inclusion (PFS2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent 1.1 Study participants must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal study participant care.

   1.2 Study participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
2. Target Population 2.1. Untreated patients with multiple myeloma diagnosis to the IMWG diagnostic criteria 2.2. Subject must have documented multiple myeloma as defined by the criteria below:

   * Monoclonal plasma cells in the bone marrow ≥10% at some point in their disease history or presence of a biopsy proven plasmacytoma.
   * Measurable disease as defined by any of the following:
   * IgG multiple myeloma: Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
   * IgA, IgD, IgE, IgM multiple myeloma: serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
   * Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum Immunoglobulin kappa lambda free light chain ratio.
3. ECOG ≤2
4. Not eligible for autologous transplantation
5. Age 18 years or above
6. Reproductive Status

   * Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception and must agree to use adequate method to avoid pregnancy for 5 months (30 days plus the time required for durvalumab to undergo five half-lives) after the last dose of study drug.

     * Appropriate methods of contraception are:

       * female sterilization or tubal ligation (at least 6 weeks prior to the start of the study treatment),
       * male sterilization (at least 6 months prior to the start of the study treatment) and/or
       * a combination of a hormonal method of contraception with a barrier method or/and
       * an intrauterine device or system
   * Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of β-HCG) within one until two weeks prior to the start of durvalumab at time of neoadjuvant treatment and after surgery before starting adjuvant treatment.
   * Women will be not be considered to be of childbearing potential if they are post-menopausal and/or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). To be considered post-menopausal the appropriate age-specific requirements have to be met:
   * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
   * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago.
   * Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving durvalumab and who are sexually active with WOCBP must be willing to adhere to contraception for a period of 7 month post treatment completion.

Exclusion Criteria:

* Subject has received any multiple myeloma therapy previously except dexamethasone to a maximum cumulative dose of 160mg, emergency radiotherapy or surgery for symptom control
* Participation in other interventional clinial trials
* Subject has known meningeal involvement of multiple myeloma.
* Subject has a history of malignancy (other than multiple myeloma) within 3 years before the date of Screening.

Subject has either of the following:

1. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 is <50% of predicted normal.
2. Known moderate or severe persistent asthma, within the past 2 years, uncontrolled asthma of any classification. Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.

   * Use of drugs with significant interaction with or intolerance to the investigational product
   * Subject is known to be seropositive for human immunodeficiency virus (HIV)
   * active hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] or positive HBV DNA)
   * Subject has any concurrent medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
   * Patients has known current symptomatic congestive heart failure (New York Heart Association Class III-IV), unstable angina pectoris, or cardiac arrhythmia
   * Subject has any of the following laboratory test results during the Screening Phase:

     * Absolute neutrophil count ≤1.0 × 109/L;
     * Platelet count <50 × 109/L
     * Aspartate aminotransferase (AST) or alanine aminotransferase level (ALT) ≥2.5 times the upper limit of normal (ULN)
     * Alkaline phosphatase level ≥2.5 × ULN
     * Total bilirubin level ≥1.5 × ULN, (except for Gilbert Syndrome: direct bilirubin 1.5 × ULN)
   * Pregnant women and nursing mothers, or a women who is planning to become pregnant while enrolled in this study or within 3 month after the last dose of daratumumab
   * Failure to use highly-effective contraceptive methods. The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly-effective:

     * Oral hormonal contraception ('pill')
     * Dermal hormonal contraception
     * Vaginal hormonal contraception (NuvaRing®)
     * Contraceptive plaster
     * Long-acting injectable contraceptives
     * Implants that release progesterone (Implanon®)
     * Tubal ligation (female sterilisation)
     * Intrauterine devices that release hormones (hormone spiral)
     * Double barrier methods This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).
   * Persons with any kind of dependency on the principal investigator or employed by the sponsor or principal investigator
   * Legally incapictated persons
   * Subject is known or suspected of not being able to comply with the study protocol(eg, because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
   * Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of induction therapy with daratumumab, bortezomib, cyclophosphamide and dexamethasone (DVCd) | 24 weeks
  Proportion of patients achieving a very good partial remission (VGPR) or better after 8 cycles of DVCd

SECONDARY OUTCOMES:
Assessment of the efficacy of maintenance therapy until progression using daratumumab in combination with bortezomib and dexamethasone. | open
  Proportion of patients with no detectable minimal residual disease as best response to maintenance therapy using daratumumab in combination with bortezomib and dexamethasone
Assessment of the efficacy of a daratumumab-containing regimen at first relapse, following a daratumumab-containing first line regimen. | up to 48 months (from first progression/relapse until second progression/relapse or death, whichever occurs first (PFS-R)
  Progression free survival from first relapse (PFS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Christof Scheid, Prof. Dr., Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No